CLINICAL TRIAL: NCT04443153
Title: Adapting Diabetes Treatment Expert Systems to Patient's Expectations and Psychobehavioral Characteristics in Type 1 Diabetes
Brief Title: Adapting Diabetes Treatment Expert Systems to Patient in Type 1 Diabetes
Acronym: DSS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marc Breton, Associate Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200007; 2R01DK051562-19A1 (NIH)
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Behavior; Continuous Glucose Monitor (CGM); Insulin Pump; Decision Support System (DSS); Personalized Feedback (PF); Sensor Augmented Pump therapy (SAP); Multiple Daily Injections (MDI); Sensor Augmented Mode (SAM); Continuous Subcutaneous Insulin Infusion (CSII)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- De-escalation (Experimental): Subjects randomized to this arm will proceed from DSS to PF to SAM
  Interventions: Device: Personalized Feedback; Device: Decision Support System; Device: Sensor Augmented Mode
- Escalation (Experimental): Subjects randomized to this arm will proceed from SAM to PF to DSS
  Interventions: Device: Personalized Feedback; Device: Decision Support System; Device: Sensor Augmented Mode

INTERVENTIONS:
Device: Personalized Feedback — Provides tailored information to the user about what glycemic risk they may be facing as well as how glycemic control and system use looked in the past week. Treatment decision and therapy changes are entirely left to the decision of the user.
Device: Decision Support System — CGM-based system that includes Personalized Feedback (PF) and further assists with treatment recommendations for common metabolic challenges
Device: Sensor Augmented Mode — A mode in Diabetes Assistant (DiAs) that combines Diabetes Assistant, Insulin pump or Multiple Daily Injections, CGM, ketone meters, and glycemic treatment guidelines together to manage diabetes.

SUMMARY:
This study is evaluate the superior efficacy of a Continuous Glucose Monitor (CGM)-based advisory system in Type 1 Diabetes Mellitus (T1DM), as compared to Sensor Augmented Mode (SAM) therapy, and with characterizing the impact of psycho-behavioral factors on system performance, which will enable system individualization and lead to automated adaptation of advice delivery to optimize glycemic control and reduce the system's psychological impact.

DETAILED DESCRIPTION:
Four cohorts of about 25 participants each (expected retention 20 per cohort). Each cohort will continue for ~7 months. Following recruitment, screening, and a run-in period of SAM, participants will be randomized into one of two groups: escalation vs. de-escalation of devices and function. Each treatment modality (SAM - Sensor-Augmented Mode, PF - Personalized Feedback, DSS - Decision Support Systems) will continue for about 8 weeks, with the last 4 weeks used to assess glucose variability (GV) from CGM data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least one year
* HbA1c 6.0-11.0%, inclusive
* Demonstration of proper mental status and cognition for the study
* If on a non-insulin hyperglycemic therapy, stability on that therapy for the prior 3 months and willingness not to alter the therapy for the study duration.
* For females, not currently known to be pregnant
* If female and sexually active, must agree to use a highly effective form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study. Also, subjects who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
* Subjects must have Internet access and a computer system that meets the requirements for uploading the study equipment and ability to participate in video conferencing.
* Investigator has confidence that the subject can successfully operate all study devices and is capable of adhering to the protocol

Exclusion Criteria:

* NPH (neutral protamine hagedorn) insulin
* Use of any medication that at the discretion of the investigator is deemed to interfere with the trial.
* Current treatment of a primary seizure disorder
* Coronary artery disease or heart failure, unless written clearance is received from a cardiologist.
* Hemophilia or any other bleeding disorder
* A known medical condition, which in the opinion of the investigator or designee, would put the participant or study at risk such as the following examples:

  * Inpatient psychiatric treatment in the past 6 months
  * Presence of a known adrenal disorder
  * Abnormal liver function test results (Transaminase >3 times the upper limit of normal)
  * Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2).
  * Active gastroparesis requiring medical therapy
  * Uncontrolled thyroid disease (TSH undetectable or >10 mlU/L).
  * Abuse of alcohol or recreational drugs
  * Infectious process not anticipated to be resolved prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis, deep tissue infection).
  * Uncontrolled arterial hypertension (Resting diastolic blood pressure >100 mmHg and/or systolic blood pressure >180 mmHg).
  * Uncontrolled microvascular complications such as current active proliferative diabetic retinopathy defined as proliferative retinopathy requiring treatment (e.g. laser therapy or VEGF inhibitor injections) in the past 12 months.
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol.
* Not familiar with smart phone technology
* Current use of the following drugs and supplements:

  * Oral steroids
  * Any other medication that the investigator believes is a contraindication to the subject's participation
* Participation in another pharmaceutical or device trial at the time of enrollment or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Breton, PhD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Pending

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment began September 4, 2020, and all study activities were completed on September 19, 2024. As defined in the protocol, a participant is considered enrolled when the informed consent form has been signed by the participant and the study team. Eighty-eight (88) signed consent, and 26 participants screen failed, withdrew, or dropped prior to screening.
Pre-assignment Details: Once eligibility and device training was completed, participants completed a minimum of 14 days (if CGM use within the preceding 3 months) or 4 weeks (if no CGM use within the preceding 3 months) of home use of the DiAs system in Sensor-Augmented Mode (SAM). One participant elected to withdraw from the study.
Period: First intervention (8 weeks)
Arm/Group | Escalation | De-escalation
Started | 32 | 29
Completed | 30 | 27
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 2
Period: Second intervention (8 weeks)
Arm/Group | Escalation | De-escalation
Started | 30 | 27
Completed | 27 | 26
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Period: Third Intervention (8 weeks)
Arm/Group | Escalation | De-escalation
Started | 27 | 26
Completed | 27 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escalation | De-escalation | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (11.1) | 36.9 (12.7) | 37.3 (11.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 11 | 13 | 24
  Gender: Female | 16 | 12 | 28
  Gender: Prefer not to say | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 25 | 51
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Highest education level [Count of Participants; unit: Participants]
  High school degree or equivalent (e.g., GED) | 4 | 4 | 8
  Some college but no degree | 2 | 5 | 7
  Associate degree | 5 | 2 | 7
  Bachelor degree | 11 | 8 | 19
  Graduate degree | 5 | 7 | 12
Last year household income [Count of Participants; unit: Participants]
  Less than $20,000 | 1 | 0 | 1
  $20,000 - $44,999 | 1 | 2 | 3
  $45,000 - $99,999 | 15 | 12 | 27
  $100,000 - $149,999 | 4 | 8 | 12
  $150,000 - $199,999 | 3 | 2 | 5
  More than $200,000 | 1 | 1 | 2
  Prefer not to answer | 2 | 1 | 3
Health Insurance [Count of Participants; unit: Participants]
  Private insurance through my employer | 19 | 16 | 35
  Self-insured with private health insurance | 3 | 2 | 5
  Public state or federal health insurance (Medicaid, Medicare, Veteran's Health Affairs...) | 3 | 6 | 9
  Uninsured | 2 | 1 | 3
  Prefer not to answer | 0 | 1 | 1
Number of participants with each infusion set type [Count of Participants; unit: Participants]
  MDI | 18 | 14 | 32
  Pump | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Outcomes
Description: Glucose Variability (GV) as measured by CGM-based Coefficient of Variation (CV), as recommended by the International Consensus on Use of Continuous Glucose Monitoring.
Time Frame: Assessed over the last 4 weeks (Weeks 4 - 8), for each intervention
Measure: Mean (Standard Deviation); unit: Percent of coefficient of variation
Arm/Group | Escalation | De-escalation
Number analyzed (Participants) | 27 | 26
Percent of coefficient of variation
  SAM | 36.3 (4.0) | 35.7 (6.7)
  PF | 37.5 (5.3) | 35.8 (6.0)
  DSS | 38.6 (5.1) | 35.8 (6.6)

2. Secondary Outcome: Percent Time in Clinical Hypoglycemia
Description: Percentage of time blood glucose was below 54mg/dL as per CGM
Time Frame: Assessed over the last 4 weeks (Weeks 4 - 8), for each intervention
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Escalation | De-escalation
Number analyzed (Participants) | 27 | 26
Percent of time
  SAM | 0.5 (0.8) | 0.7 (0.7)
  PF | 0.6 (0.6) | 0.6 (1.0)
  DSS | 0.7 (0.9) | 0.6 (0.9)

3. Secondary Outcome: Percent Time Below Recommended Threshold
Description: Percentage of time blood glucose was below 70mg/dL as per CGM
Time Frame: Assessed over the last 4 weeks (Weeks 4 - 8), for each intervention
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Escalation | De-escalation
Number analyzed (Participants) | 27 | 26
Percentage of time
  SAM | 2.5 (2.4) | 3.5 (3.3)
  PF | 3.1 (2.6) | 2.8 (2.9)
  DSS | 2.8 (2.3) | 2.9 (2.9)

4. Secondary Outcome: Percent Time in Target Range
Description: Percentage of time blood glucose was 70mg/dL and 180mg/dL as per CGM
Time Frame: Assessed over the last 4 weeks (Weeks 4 - 8), for each intervention
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Escalation | De-escalation
Number analyzed (Participants) | 27 | 26
Percentage of time
  SAM | 53.9 (16.9) | 60.1 (16.9)
  PF | 53.6 (18.3) | 61.1 (16.1)
  DSS | 53.3 (16.0) | 57.5 (15.8)

5. Secondary Outcome: Percent Time Above Range
Description: Percentage of time blood glucose was above 180mg/dL as per CGM
Time Frame: Assessed over the last 4 weeks (Weeks 4 - 8), for each intervention
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Escalation | De-escalation
Number analyzed (Participants) | 27 | 26
Percent of time
  SAM | 43.6 (18.2) | 36.4 (18.8)
  PF | 43.3 (19.7) | 36.1 (17.4)
  DSS | 43.9 (16.7) | 39.6 (16.6)

6. Secondary Outcome: Percent Time Above 250 mg/dL
Description: Percentage of time blood glucose was above 250mg/dL as per CGM
Time Frame: Assessed over the last 4 weeks (Weeks 4 - 8), for each intervention
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Escalation | De-escalation
Number analyzed (Participants) | 27 | 26
Percentage of time
  SAM | 16.6 (12.6) | 11.4 (11.0)
  PF | 18.4 (14.5) | 12.2 (12.0)
  DSS | 19.4 (14.8) | 13.3 (11.5)

7. Secondary Outcome: Average Glycemia
Description: average of CGM values
Time Frame: Assessed over the last 4 weeks (Weeks 4 - 8), for each intervention
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Escalation | De-escalation
Number analyzed (Participants) | 27 | 26
mg/dl
  SAM | 179.1 (32.3) | 164.9 (31.2)
  PF | 179.8 (35.5) | 167.3 (30.6)
  DSS | 182.2 (33.0) | 172.2 (27.5)

8. Secondary Outcome: Low Blood Glucose Index
Description: The low blood glucose index (LBGI) is based on a nonlinear transformation of blood glucose values that corrects for the asymmetry of the glucose scale. This transformation maps glucose values into a risk space (minimum risk = 0), where higher values correspond to higher risk. Values <1 suggest low risk of hypoglycemia.
Time Frame: Assessed over the last 4 weeks (Weeks 4 - 8), for each intervention
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Escalation | De-escalation
Number analyzed (Participants) | 27 | 26
index
  SAM | 0.7 (0.5) | 0.9 (0.7)
  PF | 0.8 (0.6) | 0.8 (0.7)
  DSS | 0.8 (0.5) | 0.7 (0.6)

9. Secondary Outcome: High Blood Glucose Index
Description: The high blood glucose index (HBGI) is based on a nonlinear transformation of blood glucose values that corrects for the asymmetry of the glucose scale. This transformation maps glucose values into a risk space (minimum risk = 0), where higher values correspond to higher risk. Values below 10 suggest low to moderate risk.
Time Frame: Assessed over the last 4 weeks (Weeks 4 - 8), for each intervention
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Escalation | De-escalation
Number analyzed (Participants) | 27 | 26
index
  SAM | 10.6 (5.7) | 8.3 (5.0)
  PF | 11.0 (6.2) | 8.7 (5.3)
  DSS | 11.4 (6.2) | 9.4 (4.8)

ADVERSE EVENTS:
Time Frame: 7 months
Description: Adverse Event definitions are the same as ClinicalTrials.Gov. Please see protocol for further details about adverse event reporting.
Groups:
- Sensor-augmented mode (SAM): Sensor Augmented Mode: A mode in Diabetes Assistant (DiAs) that combines Diabetes Assistant, Insulin pump or Multiple Daily Injections, CGM, ketone meters, and glycemic treatment guidelines together to manage diabetes.
- Personalized Feedback (PF): Personalized Feedback: Provides tailored information to the user about what glycemic risk they may be facing as well as how glycemic control and system use looked in the past week. Treatment decision and therapy changes are entirely left to the decision of the user.
- Decision support system (DSS): Decision Support System: CGM-based system that includes Personalized Feedback (PF) and further assists with treatment recommendations for common metabolic challenges
Arm/Group | Sensor-augmented mode (SAM) | Personalized Feedback (PF) | Decision support system (DSS)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/53 | 1/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensor-augmented mode (SAM) (N=53) | Personalized Feedback (PF) (N=53) | Decision support system (DSS) (N=53)
Severe Hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) — High BGs night before event. BG=340 @645 AM-took Humalog 3u & Lantus 6u @730 AM. BG=68 at 8 AM-Took 100g carbs. BG=280 @10 AM-took Humalog 2u. Very active in AM. Seizure ~1130 AM. CGM=66 @1135 AM. EMS glucose tx. Fully recovered/no hospitalization.
Severe Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) — Woke by alarm @4:45 AM. CGM=100mg/dL trending down; intent to sleep 15 min. Wellness check at 830AM when he didn't respond to spouse's call-drank juice provided by friend. CGM=42mg/dL @850AM. At 9:00 AM, participant reports feeling better.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT04443153/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT04443153/ICF_000.pdf